CLINICAL TRIAL: NCT04394650
Title: A Phase I, Multi Center, Open Label Study of CC-98633, BCMA Targeted NEX-T Chimeric Antigen Receptor (CAR) T Cells, in Subjects With Relapsed and/or Refractory Multiple Myeloma
Brief Title: A Study of CC-98633, BCMA-targeted Chimeric Antigen Receptor (CAR) T Cells, in Participants With Relapsed and/or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Juno Therapeutics, a Subsidiary of Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-98633-MM-001; U1111-1251-3435 (Other: WHO)
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Myeloma; Myeloma Multiple; CC-98633; BCMA; CAR-T; CART; BCMA CART; BCMA CAR-T
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CC-98633 (Experimental): Subjects will receive CC-98633 following 3 consecutive doses of lymphodepleting chemotherapy (fludarabine and cyclophosphamide).
  Interventions: Biological: CC-98633

INTERVENTIONS:
Biological: CC-98633 — Subjects will undergo leukapheresis to isolate peripheral blood mononuclear cells (PBMCs) to produce CC-98633.
  During CC-98633 production, subjects may receive bridging chemotherapy for disease control. Upon successful generation of CC-98633 product, subjects will receive treatment with CC-98633 therapy.
  Study treatment will include lymphodepleting chemotherapy followed by one dose of CC-98633 administered by intravenous (IV) injection.

SUMMARY:
This is a Phase 1, multicenter, open-label study of CC-98633, BCMA-Targeted NEX-T Chimeric Antigen Receptor (CAR) T Cells, in participants with relapsed and/or refractory multiple myeloma.

The study will consist of 2 parts: dose-escalation (Part A) and dose-expansion (Part B). The dose-escalation part (Part A) of the study is to evaluate the safety and tolerability of increasing dose levels of CC-98633 to establish a recommended Phase 2 dose RP2D(s); and the dose-expansion part (Part B) of the study is to further evaluate the safety, pharmacokinetics/pharmacodynamics, and efficacy of CC-98633 at the RP2D(s).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Signed written informed consent prior to any study procedure.
3. Relapsed and/or refractory multiple myeloma (MM).

   1. Subjects must have documented progressive disease as per International Myeloma Working Group (IMWG) criteria during or within 12 months of completing treatment with the last anti-myeloma treatment regimen before study entry. Also, subjects with confirmed progressive disease within 6 months prior to start of Screening and who are refractory (or non-responsive) to their most recent anti-myeloma treatment regimen afterwards will be also eligible.
   2. Part A and Part B Cohort A: Subjects must have confirmed at least 3 prior antimyeloma treatment regimens.
   3. Part B Cohort B only: Subjects must have received at least 1 but no greater than 3 prior antimyeloma treatment regimens, including a proteasome inhibitor and immunomodulatory agent.
   4. Subjects must have previously received all of the following therapies:

   i) Autologous stem cell transplant ii) A regimen that included an immunomodulatory agent (eg, thalidomide, lenalidomide, pomalidomide) and a proteasome inhibitor (eg, bortezomib, carfilzomib, ixazomib), either alone or combination iii) Anti-CD38 (eg, daratumumab), either alone or combination Subjects in Cohort B do not require prior anti-CD38 antibody therapy.
4. Measurable disease
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
6. Adequate organ function

Exclusion Criteria:

1. Known active or history of central nervous system (CNS) involvement of MM
2. Active or history of plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, skin changes) syndrome, or clinically significant amyloidosis
3. Prior treatment with CAR T-cell or another genetically modified T-cell therapy
4. Part A and Part B Cohort A only: Prior treatment with investigational therapy directed at BCMA
5. Uncontrolled or active infection
6. Active autoimmune disease requiring immunosuppressive therapy
7. History or presence of clinically significant CNS pathology such as seizure disorder, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | From the time of informed consent and follow up to 2 years after infusion of CC-98633:
  incidence and severity of AEs. An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 2 years after CC-98633 infusion
  The proportion of subjects with a partial response (PR) or better by the IMWG criteria.
Complete Response (CR) Rate | Up to 2 years after CC-99633 infusion
  The proportion of subjects achieving stringent CR or CR.
Duration of response (DOR) | Up to 2 years after CC-98633 infusion
  The time from first response (sCR, CR, VGPR, or PR) to progressive disease (PD) or death.
Time to response (TTR) | Up to 2 years after CC-98633 infusion
  Time from CC-98633 infusion to the first documentation of response (sCR, CR, VGPR or PR).
Time to complete response (TTCR) | Up to 2 years after CC-98633 infusion
  Time from CC-98633 infusion to the first documentation of sCR or CR
Progression free survival (PFS) | Up to 2 years after CC-98633 infusion
  Time from CC-98633 infusion to the first documentation of PD, or death from any cause, whichever occurs first
Overall survival (OS) | Up to 2 years after CC-98633 infusion
  Time from CC-98633 infusion to death
Pharmacokinetics - maximum serum concentration (Cmax) | Up to 2 years after CC-98633 infusion
  Maximum blood concentration
Pharmacokinetics -time to peak serum concentration (tmax) | Up to 2 years after CC-98633 infusion
  Time to peak (maximum) blood concentration
Pharmacokinetics - Area under curve (AUC) | Up to 2 years after CC-98633 infusion
  Area under the curve
Very good partial response (VGPR) or better | Up to 2 years after CC-98633 infusion
  Is define as proportion of subjects achieving sCR, CR, or VGPR

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (11):
- United States (11):
  - Local Institution - 103, Birmingham, Alabama
  - Local Institution - 111, Phoenix, Arizona
  - Local Institution - 110, Stanford, California
  - Local Institution - 107, Chicago, Illinois
  - Local Institution - 101, Westwood, Kansas
  - Local Institution - 109, Rochester, Minnesota
  - Local Institution - 106, Buffalo, New York
  - Local Institution - 104, New York, New York
  - Local Institution - 102, New York, New York
  - Local Institution - 108, Charlotte, North Carolina
  - Local Institution - 105, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/content/studyconnect/us/en/clinical-trials/NCT04394650.html